CLINICAL TRIAL: NCT03238248
Title: A Phase II Trial of Pevonedistat and Azacitidine in MDS or MDS/MPN Patients Who Fail Primary Therapy With DNA Methyl Transferase Inhibitors
Brief Title: Pevonedistat and Azacitidine in MDS or MDS/MPN Patients Who Fail Primary Therapy With DNA Methyl Transferase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sanjay Mohan, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HEM 16146; NCI-2017-01377 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Myelodysplastic Syndromes; Myeloproliferative Neoplasm
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pevonedistat and Azacitidine (Experimental): Participants will receive Azacitidine (via an injection under the skin, or via an intravenous infusion (IV bag) on days 1, 2, 3, 4 and 5 of each 28-day cycle.
  Participants will receive Pevonedistat (through a vein in the arm) on Days 1, 3 and 5 of each 28-day cycle.
  Interventions: Drug: Azacitidine Subcutaneous Injection or Intravenous Infusion; Drug: Pevonedistat Infusion; Procedure: Bone Marrow Biopsy & Aspirate

INTERVENTIONS:
Drug: Azacitidine Subcutaneous Injection or Intravenous Infusion — 75 mg/m2
Drug: Pevonedistat Infusion — 20 mg/m2
Procedure: Bone Marrow Biopsy & Aspirate — Removal of a small piece of bone and bone marrow by inserting a needle into hip bone.

SUMMARY:
This study will evaluate the treatment combination of pevonedistat and azacitidine in the setting of DNA methyltransferase inhibitor(s) failure in patients with relapsed/refractory myelodysplastic syndrome or myelodysplastic syndrome/myeloproliferative neoplasm.

DETAILED DESCRIPTION:
Primary Objective:

To compare survival of patients treated with a combination of pevonedistat and azacitidine after failure of DNA methyltransferase inhibitors (DNMTi) to historical survival for patients with relapsed/refractory myelodysplastic syndrome (MDS) or myelodysplastic/ myeloproliferative overlap syndromes (MDS/MPN) who are ineligible for hematopoietic stem cell transplant (HSCT)

Secondary Objectives:

* To determine the rate of hematologic improvement (HI) in patients with relapsed/refractory MDS or MDS/MPN treated with pevonedistat and azacitidine after DNMTi failure
* To determine the complete remission (CR) and marrow CR rates in patients with relapsed/refractory MDS or MDS/MPN treated with pevonedistat and azacitidine after DNMTi failure
* To determine the reduction of bone marrow blasts in patients with relapsed/refractory MDS or MDS/MPN treated with pevonedistat and azacitidine after DNMTi failure

Exploratory Objectives:

* To correlate the mutation burden in patients with relapsed/refractory MDS or MDS/MPN with response to treatment with pevonedistat and azacitidine
* To correlate genomic aberrations with rate of response and survival in relapsed/refractory MDS or MDS/MPN patients treated with pevonedistat and azacitidine
* To measure the effect of pevonedistat treatment in combination with azacitidine on quality of life in patients with relapsed/refractory MDS or MDS/MPN
* To define epigenetic biomarkers for pevonedistat use in relapsed/refractory MDS or MDS/MPN

ELIGIBILITY:
Inclusion:

* Signed and dated voluntary written informed consent before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* Male or female ≥ 18 years of age.
* Morphologically confirmed diagnosis of MDS or MDS/MPN in accordance with WHO diagnostic criteria.
* ECOG performance status of 0, 1 or 2.
* Expected survival ≥ 3 months after consenting.
* Refractory/relapsed disease following DNMTi failure. Refractory disease defined as either:

  * failure to achieve an objective response after at least 4 cycles of DNMTi therapy, or
  * failure to achieve an objective response with clear progressive disease on bone marrow biopsy after at least 2 cycles of DNMTi therapy. Relapsed disease is defined as having progressive disease after achieving an objective response after at least 2 cycles of DNMTi therapy.

Previous DNMTi therapy may include 5'azacitidine, decitabine, or DNMTi therapy currently in clinical trials (e.g. SGI-110 (guadecitabine), ASTX727 or CC-486).To be considered DNMTi treatment failure, during each prior treatment cycle, patients must have received equivalent to minimum dosing of:

decitabine 15mg/m2 daily x 5 days, or

5'azacitidine 50mg/m2 IV/SC daily x 5 days,

SGI-110 (guadecitabine) 60mg/m2 SC daily x 5 days, or

oral DNMTi therapy with ASTX727 20/100mg daily x 5 days, or

oral DNMTi therapy with CC-486 200mg daily x 14 days

* Recovery to ≤ Grade 1 or baseline of any toxicity due to prior systemic treatments, excluding alopecia.
* Patient consent to collection of fresh bone marrow biopsy and aspirate for exploratory research obtained from a procedure performed no more than 28 days prior to initiating treatment on Cycle 1, Day 1. Requirement for bone marrow biopsy may be waived with approval of the study chair in the event that a bone marrow biopsy cannot be obtained.
* Clinical laboratory values as specified below:

  * Serum albumin > 2.7 g/dL
  * Total bilirubin ≤ 1.5 x ULN
  * ALT and AST ≤ 2 x ULN
  * Calculated creatinine clearance ≥ 50 mL/min (per the Cockcroft-Gault formula)
  * WBC ≤ 50,000/µL (use of hyroxyurea is permitted)
* Hgb <8g/dL should be transfused to provide adequate tissue perfusion as per the discretion of the investigators and local practice. Rechecking Hgb level prior to start on Cycle 1 Day 1 is not necessary as long as patients do not have inadequate oxygenation, underlying cardiopulmonary compromise, and/or any other reason deemed clinically significant to delay therapy per the investigator.
* Women of childbearing potential must have a negative serum pregnancy test; and additionally agree to simultaneously use at least 2 methods of effective contraception or abstain from heterosexual intercourse from the time of signing consent, and until 4 months after patient's last dose of protocol-indicated treatment. Periodic abstinence (e.g. calendar,ovulation, symptothermal, postovulation methods for the female partner) and withdrawal are not acceptable methods of contraception.

Women of child bearing potential are defined as those not surgically sterile or not post-menopausal. If a female patient has not had a bilateral tubal ligation, a bilateral oophorectomy, or a complete hysterectomy; or has not been amenorrheic for at least 1 year in the absence of an alternative medical cause, then patient will be considered a female of childbearing potential. Postmenopausal status in females under 55 years of age should be confirmed with a serum FSH level within laboratory reference range for postmenopausal women.

- Men, even if surgically sterilized (i.e. status post-vasectomy), who are sexually active with women of childbearing potential must agree to follow instructions for effective barrier contraception from the time of signing consent and until 4 months after last dose of protocol-indicated treatment. Periodic abstinence (e.g. calendar, ovulation, symptothermal, postovulation methods for the female partner) and withdrawal are not acceptable methods of contraception.

Exclusion:

* Diagnosis of acute myeloid leukemia (i.e. ≥ 20% peripheral or marrow blasts).
* Any HSCT within 6 months prior to signing informed consent.
* Any patient who is eligible for HSCT at the time of study screening.
* Clinically significant graft versus host disease (GVHD) or GVHD requiring initiation of treatment or treatment escalation within 21 days, and/or > Grade 1 persistent or clinically significant non-hematologic toxicity related to HSCT
* Any previous treatment with pevonedistat or other NEDD8 inhibitor.
* Treatment with any investigational products within 14 days before the first dose of protocol-indicated treatment.
* Systemic antineoplastic therapy or radiotherapy within 14 days before the first dose of any study drug.
* Major surgery requiring general anesthesia within 14 days before the first dose of any study drug or a scheduled surgery during study period. (Placement of a central line or port-a-catheter is acceptable within this time frame and does not exclude the patient.)
* Treatment with clinically significant metabolic CYP3A inducers within 14 days before the first dose of study drug. Clinically significant CYP3A inducers are not permitted during the study.
* Prolonged QTc interval > 500 msec, calculated according to Fredericia's formula
* Known cardiopulmonary disease defined as having one or more of the following:

  * Uncontrolled high blood pressure (i.e. systolic > 180 mmHg or diastolic > 95 mmHg);
  * Symptomatic cardiomyopathy;
  * Ischemic heart disease; Patients with acute coronary syndrome, myocardial infarction, and/or revascularization (e.g. coronary artery bypass graft, stent) within 6 months of first dose of study drug are excluded; Patients with a history of ischemic heart disease who have had revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll;
  * Arrhythmia (e.g. history of polymorphic ventricular fibrillation or torsade de pointes). Patients with symptomatic atrial fibrillation (Afib) incompletely controlled medically, or controlled by device (e.g. pacemaker) or by ablation in the past 6 months are excluded. However, patients with stable, AFib for a period of at least 6 months, whose Afib is controlled with medication, or who have a history of paroxysmal AFib are permitted to enroll;
  * Implantable cardioverter defibrillator;
  * Congestive heart failure (New York Heart Association [NYHA] Class III or IV; or Class II with a recent decompensation requiring hospitalization or referral to a heart failure clinic within 4 weeks before screening),
  * Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing). Mild regurgitation is not excluded;
  * Pulmonary hypertension.
* Female patients who are both lactating and breastfeeding, who have a positive serum pregnancy test during screening, or who plan to become pregnant while in the trial or within 90 days after receiving protocol-directed treatment.
* Active uncontrolled infection. Patients with infection under active treatment and controlled with antibiotics are not excluded.
* Known Childs class B or C hepatic cirrhosis or severe pre-existing hepatic impairment.
* Known hepatitis B surface antigen seropositivity or known or suspected active hepatitis C infection. Note: Patients who have isolated positive hepatitis B core antibody (i.e. in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load.
* Known human immunodeficiency virus (HIV) seropositivity.
* Any serious concurrent condition that could, in the investigator's opinion, significantly interfere with completion of study procedures or protocol compliance.
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mohan, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (5):
- United States (5):
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Kansas Cancer Center, Westwood, Kansas
  - Memorial Sloan-Kettering, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Pevonedistat and Azacitidine: Participants will receive Azacitidine (via an injection under the skin, or via an intravenous infusion (IV bag) on days 1, 2, 3, 4 and 5 of each 28-day cycle.
  Participants will receive Pevonedistat (through a vein in the arm) on Days 1, 3 and 5 of each 28-day cycle.
  Azacitidine Subcutaneous Injection or Intravenous Infusion: 75 mg/m2
  Pevonedistat Infusion: 20 mg/m2
  Bone Marrow Biopsy & Aspirate: Removal of a small piece of bone and bone marrow by inserting a needle into hip bone.
Period: Overall Study
Arm/Group | Pevonedistat and Azacitidine
Started | 71
Completed | 4
Not Completed | 67
Not completed — Death | 5
Not completed — Withdrawal by Subject | 7
Not completed — Participant proceeding to transplant | 10
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 3
Not completed — Transitioning to another study | 1
Not completed — No longer benefiting | 1
Not completed — Other complicating disease | 1
Not completed — Adverse Event | 5
Not completed — Disease progression | 26
Not completed — N/A participant is still on treatment | 1
Not completed — Decline in condition | 1
Not completed — Alternative therapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 62
  More than one race | 1
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Overall Survial Time
Description: Overall survival time is defined as time from day 1 in cycle 1 to death for any reason. Patiens alive at last follow up were censored. Overall survival time will be summarized using the method of Kaplan and Meier.
Time Frame: up to 2 years after treatment, a maximum possible duration of 38 months.
Population: Patients diagnosed with MDS or MDS/MPN and received treatment. Excluded one patient who did not start the thearpy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 70
months | 18.3 [14.4 to 30.9]

2. Secondary Outcome: Time to Progression
Description: Progression-free survival time is defined as time from day1 in cycle 1 to progression or death. Those alive without progression at the last follow up were censored. This survival will be summarized using the method of Kaplan and Meier.
Time Frame: Up to 24 months, or death
Population: Patients diagnosed with MDS or MDS/MPN and received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 70
months | 9.9 [6.0 to 17.5]

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as the percentage of patients with best response of Complete remission (CR), Hematologic improvement (HI), Marrow CR (mCR), or Partial remission (PR) among all patients evaluated. The other categories of response are progressive disease, stable disease and inevaluable. The modified recommendations of the International Working Group (IWG) for Response Criteria for altering natural history of MDS , as well as the International Consortium of clinical experts in MDS/MPN devised uniform response criteria and criteria for disease progression in MDS/MPN overlap syndromes based on three independent academic MDS/MPN workshops (Marsh 2013, December 2013 and June 2014) were used for response assessment.
Time Frame: Up to 12 months
Population: Patients with MDS or MDS/MPN received treatment and had been evaluated for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 67
percentage of participants | 23.9 [15.3 to 35.3]

4. Secondary Outcome: Rate of Hematologic Response Per IWG
Description: Will assess complete and differential blood counts (peripheral blood), and transfusion requirements. The rate of hematologic improvement is defined as the percentage of patients with only hematologic improvement (defined in the protocol) among all patients evaluated for response.
Time Frame: Up to 24 months
Population: MDS or MDS/MPN patients received treatment and evaluated for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 67
percentage of participants | 7.5 [3.2 to 16.3]

5. Other Pre Specified Outcome: Rate of Marrow Complete Response (mCR)
Description: Will assess morphologic features (e.g. presence of dysplastic features), presence of cytogenetic and/or molecular aberrancies, and myeloblast count. mCR is defined as the percentage of patients with only marrow CR among all patients evaluated.
Time Frame: Up to 24 months.
Population: MDS or MDS/MPN patients received treatment and evaluated for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 67
percentage of participants | 11.9 [6.2 to 21.8]

6. Other Pre Specified Outcome: Change in Number of Mutations as Assessed by Next Generation Sequencing (NGS)
Description: Number of specific molecular mutations in a NGS panel of 37 genes frequently mutated in myeloid malignancies will be determined by next generation sequencing before and after protocol-directed therapy. Results will be correlated with response. Clonal evolution and the relationship between response rates and mutations will be explored.
Time Frame: Up to 24 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Allele Frequency Assessed by Next Generation Sequencing (NGS)
Description: Allele frequency of specific molecular mutations in a NGS panel of 37 genes frequently mutated in myeloid malignancies will be determined by next generation sequencing before and after protocol-directed therapy. Results will be correlated with response. Clonal evolution and the relationship between response rates and mutations will be explored.
Time Frame: Up to 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious and other (not including serious) adverse events were assessed from initiation of investigational treatment (to also include events preceding initiation of study) through 30 days after last dose of investigational treatment up to a maximum duration of 2 years. All-Cause Mortality was assessed up to 38 months.
Arm/Group | Pevonedistat and Azacitidine
All-Cause Mortality (participants affected / at risk) | 49/71
Serious Adverse Events (participants affected / at risk) | 29/71
Other Adverse Events (participants affected / at risk) | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pevonedistat and Azacitidine (N=71)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 (9)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Allergic reaction (Immune system disorders) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Pancytopenia (Investigations) | 1 (1)
Pseudomonas Bacteremia (Infections and infestations) | 1 (1)
Left Hip Cellulitis (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Alkaline phosphatase Increased (Investigations) | 1 (1)
Aspartate aminotransferase Increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (6)
Hemorrhagic metastatic disease (Nervous system disorders) | 1 (1)
Face infection (Infections and infestations) | 1 (1)
Labia infection (Infections and infestations) | 1 (1)
Thromboembolic event - Related to vascular access device removal (Vascular disorders) | 1 (1)
Seronegative inflammatory migratory arthritis (General disorders) | 1 (1)
Facial Cellulitis (Infections and infestations) | 1 (1)
Suprapubic cellulitis (Infections and infestations) | 1 (1)
C.Diff Diarrhea, positive GI panel (Gastrointestinal disorders) | 1 (1)
Dental abscesses (General disorders) | 1 (1)
Acute febrile neutrophillic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Progressive disease (General disorders) | 1 (1)
Enlarged spleen (Blood and lymphatic system disorders) | 1 (1)
Peri-rectal Abscess (Gastrointestinal disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Cortical Laminar Necrosis (Nervous system disorders) | 1 (1)
Multiple Chronic Infarcts (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT03238248/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03238248/ICF_000.pdf